CLINICAL TRIAL: NCT06903780
Title: A Retrospective Survey Of The Time Course And Nature Of The Experience Of Initiating Biologic Treatment For People With Severe Asthma.
Brief Title: Experience of Biologic Treatments for Severe Asthma: a Survey
Acronym: SHARP EoB
Status: Recruiting | Type: Observational
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Plymouth (Other); University Hospital Plymouth NHS Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); University Hospital Birmingham (Other); Barts Helth NHS Trust (Unknown); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2502729; CPMS ID: 60193 (Other: NIHR Research Delivery Network (RDN))
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-11

CONDITIONS: Severe Asthma
Keywords: asthma; survey; patient perspectives; patient centred; co-development; multi-centre
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Survey using a questionnaire. — A short 23-item survey concerning patients' experiences of their biologic treatments for their severe asthma.

SUMMARY:
Severe asthma is a disease characterised by respiratory and non-respiratory symptoms. The respiratory symptoms can include breathlessness, wheeze and asthma attacks. The disease can come to dominate patients' lives, impacting their social, working and personal lives, leading to depression, anxiety and feelings of social isolation.

There are now 7 different biologic treatments available on the NHS in the UK for severe asthma. These treatments have dramatically changed how severe asthma can be treated. Research has typically focused on the benefits of these drugs from a clinical perspective, e.g., improvements in lung function, blood tests and reduction in frequency of asthma attacks and use of steroid tablets.

While these are important outcomes, they do not reflect the experiences of patients receiving these treatments, which can vary greatly. First, not all patients benefit to the same degree. Second for patients who do respond, some respond slower than others. Third while these treatments target respiratory symptoms, some patients report wider benefits, such as reductions in fatigue, depression, ability to engage in family life and other daily activities. Fourth, patients report different side effects when starting these treatments and sometimes for months afterwards, including headaches, fatigue, mental fog and joint pain. These experiences are reported by clinicians and patients, but the extent of these four variations is poorly understood, and potential reasons for them have not been explored.

To describe these differences between patients' experiences and begin understanding why they are present, we have co-designed a survey with people who have lived experience of severe asthma who are members of the European Lung Foundation's (ELF) Patient Advisory Group (PAG). This process has resulted in a survey that contains content important to patients and is worded in a way that avoids confusion regarding the meaning of the questions.

DETAILED DESCRIPTION:
A multi-centre cross-sectional survey to retrospectively assess patients' perceptions of their responses to biologic treatments for their severe asthma.

Methods A total of 400 patients will be recruited from the severe asthma centres responsible for their clinical care.

Leads from each participating site will identify patient's eligible to take part in the study. Each lead for a site will be provided with unique 'Collector IDs' (that are linked with a unique survey web URL). After receiving verbal consent from each patient, the researcher at the site will allocate the patient a 'Collector ID' and unique web URL to a survey hosted on SurveyMonkey.

On visiting the survey URL, patients will be provided with study information, provide informed consent and complete the survey information.

Participants will complete the survey without any assistance from physicians or the study staff. All survey questions and responses will be provided in the participants' native languages. All processes will be monitored by a study coordinator to assess recruitment and the completion of the survey.

Variables

Variables from the patient survey will include:

* Experience of starting a biologic treatment

  o What changed, when did the change take place and to what degree was the change experienced.
* Side effects experienced after taking a biologic treatment. Demographics
* Gender
* Age Medication use
* Use of OCS
* Use of biologic treatment Data analysis

  1. To describe the time course and nature of response in people with severe asthma who continue to be prescribed biologics for between 6 - 18 months.
* Demographics data and other survey responses will be reported as descriptive statistics including mean (SD).
* We will report a frequency distribution of responses for each survey item to describe the samples experience of biologic drugs for their severe asthma.
* To assess for the presence of recall differences between those who have been on a biologic for <12 months vs those on a biologic for ≥12 months data from these participants will be stratified and compared.

  2. To identify subgroups of response pattern to biologic treatments for severe asthma.

Analysis will be exploratory and descriptive, with relationships between survey responses identified through correlations. These correlations will provide insight into which experiences of biologic treatment (response) are related. For example, the literature anticipates that a fast response will be associated with a "better" response to biologic treatments. We will define "better" from a patient perspective, by investigating the relationship between Question 8 (Satisfaction with treatment), and time to first noticed treatment response (Question 6).

3. To describe the characteristics of the different subgroups of response pattern.

* Participants demographic data will be reported as a function of the different response patterns we identify in analysis 2.

  4. To identify a set of hypotheses driven characteristics which may predict response to biologics in future longitudinal studies for people with severe asthma, including the extra-pulmonary symptoms and side effects of treatment.
* Fatigue and other side effects from biologics may be predictors of fast response or high satisfaction with treatment.
* Correlations between the different response patterns identified in analysis 2, and questions concerning side effects and extra-pulmonary questions will be calculated. These include questions: 17, 18 and 19.
* We will also calculate correlations between the response patterns we identify in analysis 2, and the biologic the patient was prescribed.

ELIGIBILITY:
Inclusion Criteria:

Receiving a biologic treatment for at least 6 months.

• But has not been on the treatment for longer than 18 months. Note: In clinical practice, a 12-month trial of biologic treatments is needed before a decision to stop/switch treatment is made. Therefore, our inclusion criteria will capture people who are non-responders to biologic treatments.

Exclusion Criteria:

* Patients will be excluded if they are unwilling/unable to provide consent to use their data.
* Patients who have switched biologics will also be excluded.
* In the opinion of the physician responsible for the care of the patient, the patient has a condition, other than asthma which is significantly contributing to their respiratory symptoms, e.g. lung cancer, heart failure or severe COPD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient has severe asthma as defined by :
  GINA step 4 & 5 Moderate to high dose ICS and a LABA or LTRI or LAMA (theophylline)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Severe asthma biologic experience survey | 6-18 month recall
  A 23-item survey concerning the experiences of severe asthma patients who have received a biologic treatment. This survey covers many aspects of experience from:
  Degree of response Time to respond Benefits first noticed - pulmonary and extra-pulmonary Changes to other medications Side effects HRQoL improvement

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Masoli, MD, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (1):
- Royal Devon University Healthcare NHS Foundation Trust, Exeter, Devon, United Kingdom

REFERENCES:
- See also: Website with information concerning this project and other projects conducted by this team — https://www.plymouth.ac.uk/research/primarycare/severe-asthma